CLINICAL TRIAL: NCT04681781
Title: SLC13A5 Deficiency: a Prospective Natural History Study - Remote Only (International)
Brief Title: SLC13A5 Deficiency Natural History Study - Remote Only
Status: Enrolling by invitation | Type: Observational
Sponsor: TESS Research Foundation (Other)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: SLC13A5RMTNHS
Record Dates: First submitted 2020-12-18; First posted 2020-12-23 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Citrate Transporter Deficiency; Epilepsy; Rare Diseases; Movement Disorders; Genetic Disorder; SLC13A5 Deficiency; EIEE25; Kohlschutter-Tonz Syndrome (non-ROGDI); 17p13.1 Deletions Confined to SLC13A5 Gene; Citrate Transporter Disorder
Keywords: Epilepsy; Rare Disease; Movement Disorders; Genetic Disorder; Citrate Transporter Disorder; SLC13A5 Deficiency; EIEE25; Neonatal seizures; autosomal recessive
MeSH Terms: conditions — Epilepsy; Rare Diseases; Movement Disorders; Genetic Diseases, Inborn; Kohlschutter Tonz syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
SLC13A5 deficiency (Citrate Transporter Disorder, EIEE 25) is a rare genetic disorder with neurodevelopmental delays and seizure onset in the first few days of life. This natural history study is designed to address the lack of understanding of disease progression and genotype-phenotype correlation. Additionally it will help in identifying clinical endpoints for use in future clinical trials.

DETAILED DESCRIPTION:
This is a longitudinal observational study for the natural history of SLC13A5 deficiency for up to 2 years. This study does not involve any therapeutic intervention. The study includes remote visits which will be done via telephone or remote video conferencing. Translators will be available during these remote visits for non-english speaking caregivers. The initial visit will consist of collecting a detailed medical history and medical records. Prior brain imaging and available EEGs will be collected and reviewed by the study neurologist. Neuropsychological assessments will be made using Vineland Adaptive Behavior Scale version 3. Brief standardized videos recorded by the caregiver will be reviewed and scored by study personnel for movement assessment. Caregiver of ages 2 and up will be asked to complete the QOL Family Impact Module and the QOL epilepsy module. In addition to the initial visit, assessments in 1st year (every 3 months) and 2nd year (every 4 months) of enrollment will be made through remote interviews. Caregiver will be asked to maintain a seizure diary for the duration of the study to assess seizure burden. Personnel having expertise to comprehensively evaluate biological pathways that are perturbed by SLC13A5 deficiency will analyze the collected data. Improved understanding of disease pathogenesis will guide therapeutics and reveal clinical endpoints for use in future clinical trials. Identifying genotype-phenotype correlations can guide prognostication, clinical management, and genetic counseling.

ELIGIBILITY:
Inclusion Criteria:

1. Parent(s)/legal representative and/or patient must be willing and able to give informed consent/assent for participation in the study.
2. Males and females of any age are eligible for this study
3. Suspected or confirmed diagnosis of SLC13A5 deficiency with genetic variants in both SLC13A5 alleles and consistent clinical characteristics. Variants of uncertain significance in one or both alleles are acceptable if deemed good candidates by participant's primary geneticist or neurologist and study personnel.
4. Participant and caregiver must be willing to provide clinical data and participate in standardized assessments.

Exclusion Criteria:

1. The presence of a second, confirmed disorder, genetic or otherwise, affecting neurodevelopment or with other overlapping symptoms of SLC13A5 deficiency.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population will consist of children or adolescents with genetically confirmed diagnosis of SLC13A5 Deficiency and consistent clinical characteristics.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
SLC13A5 deficiency motor scale assessments. | Upto 24 months
  Caregiver will be asked to record brief standardized videos capturing the degree of disordered movements. These videos will be made and reviewed for all assessment sessions. Different movements/tasks will be assessed on different scales ranging from 0 to 8. Lesser scores represent better outcome.
Developmental assessment at baseline and longitudinally using Vineland 3 | Upto 24 months
  The Vineland Adaptive Behavior Scales, Third Edition (Vineland 3) provides a comprehensive assessment of adaptive function and has been widely used in populations with intellectual and developmental disabilities. It is validated from birth to 90 years, and scores abilities across three core and two optional domains: communication, daily living skills, socialization, and motor skills and maladaptive behaviors, respectively. Completion time for the comprehensive interview is estimated at 50 minutes when all five domains are included. Reliability and validity are widely established. Vineland 3 Adaptive Behavior Scale questionnaire will be included in the remote interviews during the initial visit for baseline assessment and followed at 6 months, 12 months and 24 months for longitudinal neuropsychological assessment
Seizure burden and semiology | Upto 24 months
  Caregiver will be asked to log number and type of seizures for the 4 weeks prior to each remote interview in a seizure tracker form. Reportable seizure types are to include: simple partial seizures (focal onset with retained awareness) WITHOUT motor signs, simple partial seizures WITH motor signs, complex partial seizures (focal onset with impaired awareness), partial (focal) seizures with secondary generalization, absences, myoclonic seizures, clonic seizures, tonic seizures, atonic seizures, and generalized tonic-clonic seizures. In addition, to assess overall change in seizure burden in 4 months between the remote interviews, Seizure Global Impression of Change (Seizure GIC) will be filled at all the remote interviews. Caregiver global impression of change will be assessed using a seven-point Likert scale. In addition, caregiver impression of change in seizure frequency and duration will be assessed using a three-point Likert scale.

SECONDARY OUTCOMES:
Caregiver Quality of Life (QOL) | Upto 24 months
  Caregiver of patients of ages 2 and up will be asked to fill questionnaires related to PedsQL Family Impact Module and PedsQL Caregiver Epilepsy Module in the initial visit and thereafter at 6 months, 12 months and 24 months. PedsQL Family Impact Module assess the impact of pediatric chronic health conditions on parents/caregiver and family by measuring parent/caregiver self-reported physical, emotional, social, and cognitive functioning, communication, and worry. The PedsQL Epilepsy Module is a 29-item measure with five scales: Impact, Cognitive, Sleep, Executive Function, and Mood/Behavior. The Impact Scale assesses how epilepsy disrupts daily activities, interacting with peers, independence, and increased disease burden due to treatment.
Sleep disturbances scale for children (SDSC) | Upto 24 months
  Caregiver will be asked to fill a one-page questionnaire to assess dependents disorders of sleep. The Sleep Disturbance Scale for Children (SDSC) is a 27-item inventory rated on a 5 point Likert-type scale. The instrument's purpose is to categorize sleep disorders in children. As well as giving an overall score the instrument uses five subdomains: disorders of initiating and maintaining sleep, sleep breathing disorders, disorders of arousal, sleep-wake transition disorders, disorders of excessive somnolence, and sleep hyperhidrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Brenda E Porter, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Lucille Packard Children's Hospital, Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The study data will be retained in the study-specific REDCap data base housed at redcap.stanford.edu. Researchers and clinicians with academic interest in SLC13A5 deficiency may be provided access to data obtained through this study. Any data shared outside of Stanford University will be done so in a coded fashion with no protected health information included and with the execution of all applicable agreements or ongoing collaborations as approved in this protocol.

REFERENCES:
- [Background] Thevenon J, Milh M, Feillet F, St-Onge J, Duffourd Y, Juge C, Roubertie A, Heron D, Mignot C, Raffo E, Isidor B, Wahlen S, Sanlaville D, Villeneuve N, Darmency-Stamboul V, Toutain A, Lefebvre M, Chouchane M, Huet F, Lafon A, de Saint Martin A, Lesca G, El Chehadeh S, Thauvin-Robinet C, Masurel-Paulet A, Odent S, Villard L, Philippe C, Faivre L, Riviere JB. Mutations in SLC13A5 cause autosomal-recessive epileptic encephalopathy with seizure onset in the first days of life. Am J Hum Genet. 2014 Jul 3;95(1):113-20. doi: 10.1016/j.ajhg.2014.06.006. PMID 24995870
- [Background] Hardies K, de Kovel CG, Weckhuysen S, Asselbergh B, Geuens T, Deconinck T, Azmi A, May P, Brilstra E, Becker F, Barisic N, Craiu D, Braun KP, Lal D, Thiele H, Schubert J, Weber Y, van 't Slot R, Nurnberg P, Balling R, Timmerman V, Lerche H, Maudsley S, Helbig I, Suls A, Koeleman BP, De Jonghe P; autosomal recessive working group of the EuroEPINOMICS RES Consortium. Recessive mutations in SLC13A5 result in a loss of citrate transport and cause neonatal epilepsy, developmental delay and teeth hypoplasia. Brain. 2015 Nov;138(Pt 11):3238-50. doi: 10.1093/brain/awv263. Epub 2015 Sep 17. PMID 26384929
- [Background] Klotz J, Porter BE, Colas C, Schlessinger A, Pajor AM. Mutations in the Na(+)/citrate cotransporter NaCT (SLC13A5) in pediatric patients with epilepsy and developmental delay. Mol Med. 2016 May 26;22:310-21. doi: 10.2119/molmed.2016.00077. PMID 27261973
- [Background] Selch S, Chafai A, Sticht H, Birkenfeld AL, Fromm MF, Konig J. Analysis of naturally occurring mutations in the human uptake transporter NaCT important for bone and brain development and energy metabolism. Sci Rep. 2018 Jul 27;8(1):11330. doi: 10.1038/s41598-018-29547-8. PMID 30054523
- [Background] Bainbridge MN, Cooney E, Miller M, Kennedy AD, Wulff JE, Donti T, Jhangiani SN, Gibbs RA, Elsea SH, Porter BE, Graham BH. Analyses of SLC13A5-epilepsy patients reveal perturbations of TCA cycle. Mol Genet Metab. 2017 Aug;121(4):314-319. doi: 10.1016/j.ymgme.2017.06.009. Epub 2017 Jun 24. PMID 28673551
- [Background] Weeke LC, Brilstra E, Braun KP, Zonneveld-Huijssoon E, Salomons GS, Koeleman BP, van Gassen KL, van Straaten HL, Craiu D, de Vries LS. Punctate white matter lesions in full-term infants with neonatal seizures associated with SLC13A5 mutations. Eur J Paediatr Neurol. 2017 Mar;21(2):396-403. doi: 10.1016/j.ejpn.2016.11.002. Epub 2016 Nov 19. PMID 27913086
- [Background] Irizarry AR, Yan G, Zeng Q, Lucchesi J, Hamang MJ, Ma YL, Rong JX. Defective enamel and bone development in sodium-dependent citrate transporter (NaCT) Slc13a5 deficient mice. PLoS One. 2017 Apr 13;12(4):e0175465. doi: 10.1371/journal.pone.0175465. eCollection 2017. PMID 28406943
- [Background] Schossig A, Bloch-Zupan A, Lussi A, Wolf NI, Raskin S, Cohen M, Giuliano F, Jurgens J, Krabichler B, Koolen DA, de Macena Sobreira NL, Maurer E, Muller-Bolla M, Penzien J, Zschocke J, Kapferer-Seebacher I. SLC13A5 is the second gene associated with Kohlschutter-Tonz syndrome. J Med Genet. 2017 Jan;54(1):54-62. doi: 10.1136/jmedgenet-2016-103988. Epub 2016 Sep 6. PMID 27600704
- [Background] Yang QZ, Spelbrink EM, Nye KL, Hsu ER, Porter BE. Epilepsy and EEG Phenotype of SLC13A5 Citrate Transporter Disorder. Child Neurol Open. 2020 Jun 8;7:2329048X20931361. doi: 10.1177/2329048X20931361. eCollection 2020 Jan-Dec. PMID 32551328